CLINICAL TRIAL: NCT00132106
Title: The Effect of a-Adrenergic Receptor Blockade on Insulin-Stimulated Forearm Glucose Uptake and Metabolism in Chronic Heart Failure
Brief Title: The Effect of Alfa-Adrenergic Receptor Blockade on Insulin-Stimulated Forearm Glucose Uptake and Metabolism in Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CHFALFA
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-08

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure | interventions — Phentolamine

INTERVENTIONS:
Drug: phentolamine

SUMMARY:
The activity of the sympathetic nervous system seems to influence the uptake (and handling) of glucose by the skeletal muscle of the forearm. Conditions in which sympathetic activity is increased seem to inhibit/reduce forearm glucose uptake. Inversely a decrease in sympathetic activity seems to increase glucose uptake. This study analyzes the effect of alfa-adrenergic receptor blockade (counteracting sympathetic influence) on insulin-stimulated forearm glucose uptake in patients with increased sympathetic activity (patients with chronic heart failure).

ELIGIBILITY:
Inclusion Criteria:

* Heart failure of at least New York Heart Association (NYHA) class II
* Left ventricular ejection fraction (LVEF) <= 40%
* Age 18-75 years

Exclusion Criteria:

* Alfa-blockers, or beta-blockers with alfa-blocking activity (carvedilol)
* Tricyclic antidepressants
* Warfarin derivatives (acetylic salicylic acid and clopidogrel are allowed)
* Hospitalisation in 6 weeks prior to the study
* Any change in medication in 6 weeks prior to the study
* Unstable angina
* Orthopnoea
* Known chronic disease of the autonomic nervous system
* Diabetes mellitus
* Oedema of the lower extremities, complicating the insertion of a venous catheter in a vein on the foot

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-08

PRIMARY OUTCOMES:
change in glucose uptake

CONTACTS AND LOCATIONS:
Overall Officials: Cees J Tack, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands